CLINICAL TRIAL: NCT04300062
Title: Tumor Rebiopsy During Progression Under Immunotherapy for Patients With Lung Cancer
Acronym: REBIMMUNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200398
Record Dates: First submitted 2020-03-02; First posted 2020-03-09 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
Keywords: lung cancer; rebiopsy; immunotherapy; progression
MeSH Terms: conditions — Lung Neoplasms; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rebiopsy (Experimental)
  Interventions: Procedure: Rebiopsy

INTERVENTIONS:
Procedure: Rebiopsy — Biopsy will be carry out with flexible bronchoscopy as usual practice under local anesthesia: under endobronchial ultrasound, punction under CT scan or ultrasonography, percutaneous pleural puncturing.

SUMMARY:
The objective of the study aims to collect tumor tissue at the moment of progression under Immune checkpoint inhibitors (ICI) in biological resources center in Ambroise Paré hospital, in order to insure later study on molecular mechanism involving the progression of NSCLC and SCLC under ICI.

The further analysis of research will be performed in the EA 4340 unity, Biomarkers and Clinical Trials in cancerology and onco-hematology, UVSQ, University of Paris-Saclay.

DETAILED DESCRIPTION:
The study will consist of creation a tumor tissue bank, all sampling will be stored in the biological resources center of Ambroise Paré hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed NSCLC or SCLC;
* Patient treated priorly by ICI and progressed under ICI;
* Have provided written informed consent for the study;
* Be >/= 18 years of age on day of signing informed consent.

Exclusion Criteria:

* Patient under guardianship or curatorship;
* Unable to provide written informed consent for the study;
* Technical impossibility to carry out tissular rebiopsy under local anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of specific histomolecular resistance | At the end of study, up to 2 years
  Banking of tumor samples at progression with immune checkpoint inhibitor (ICI) in lung cancer, to evaluate the incidence of specific histomolecular resistance mechanisms to ICI by immunohistochemistry and molecular testing.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Giroux Leprieur, MD, PhD, Principal Investigator — Service de Pneumologie et Oncologie thoracique, Hôpital Ambroise Paré, APHP
Locations (1):
- Service de Pneumologie et Oncologie thoracique, Hôpital Ambroise Paré, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giroux Leprieur E, Dumenil C, Julie C, Giraud V, Dumoulin J, Labrune S, Chinet T. Immunotherapy revolutionises non-small-cell lung cancer therapy: Results, perspectives and new challenges. Eur J Cancer. 2017 Jun;78:16-23. doi: 10.1016/j.ejca.2016.12.041. Epub 2017 Apr 11. PMID 28407528